CLINICAL TRIAL: NCT05777057
Title: Comparison Between KAVO DIAGNOdent and Digital Radiography in Occlusal Caries Detection (A Diagnostic Accuracy Study)
Brief Title: Assessing Accuracy of Kavo Diagnodent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa Mahmoud Elsayed Said, Demonstrator at the Faculty of Dentistry at Misr University for Science and Technology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ORAD 3-3-1
Record Dates: First submitted 2023-02-01; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Condition
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Extracted teeth are radiographed and examined by diagnodent and then sections are examined under light microscope
Masking Description: 2 radiologist don't know the results of diagnodent and doctor in lab also don't know the the results of diagnodent and radiograph
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Extracted teeth (Other): Extracted teeth with intial caries without cavitation is examined by diagnodent and digital imaging and then by light microscope
  Interventions: Diagnostic Test: Diagnodent

INTERVENTIONS:
Diagnostic Test: Diagnodent — using DIAGNDENT depends on the principle that when 655nm wavelength of Diode laser is irradiated on dental surface, intraoral bacteria metabolites will absorb it and then metabolites emit a red fluorescence. The dental surface will reflect this fluorescence and gives number between 0 and 99 on the screen of the DIAGNdent.

SUMMARY:
This study aims to evaluate the accuracy of kavodiagondent and compare with digital radiograph (vista scan).the gold standard is light microscope

DETAILED DESCRIPTION:
Extracted teeth with intial caries (no cavitation)will be used to detect caries. The teeth will be numbered and each of the occlusal surfaces will be measured by DIAGNOdent with a conical probe in accordance with the manufacturer's instructions. The standard value for each individual tooth will be calibrated before each measurement by measuring in a region of sound tissue. The occlusal surfaces will be carefully scanned and measured 3 times when wet, and 3 times after they had been wiped with paper tissues and exposed to air for about 2 min in room temperature. The maximum value from each measurement will be registered and the mean values of the three data under wet and dry conditions, respectively, will be calculated. After an interval of 2 weeks, the procedure will be repeated under identical conditions. All occlusal surfaces will be photographed. The sites with the highest values will be indicated in the photographs in order to identify the location for the second measurement and for subsequent sectioning for light microscope examination.

The teeth will be arranged in pairs and mounted in plaster blocks. Reproducible radiographs will be obtained. This will be done by digital radiography (vista scan sensor). The radiographs will be examined by 4 radiologists. The observers will be instructed to select one of five ratings to represent his or her level of confidence that a carious lesion was present or not in the occlusal surfaces of the teeth. The following scale was used: 1 = definitely not caries, 2 = probably not Caries, 3 = questionable, 4 = probably caries, and 5 = definitely caries.

After the laser fluorescence measurements had been completed and the digital radiographs had been exposed, the teeth will be removed from the blocks and embedded in plastic. At the sites indicated in the photographs, buccolingual sections approximately 300 µm thick will be taken perpendicular to the occlusal surfaces using a water-cooled saw. The slices will then examined under light microscope. The lesion depth will be scored on a scale from 0 to 4, where 0 = sound, 1 = enamel caries limited to the outer half of the enamel, 2 = enamel caries in the inner half of the enamel, 3 = dentinal caries in the outer half of the dentine, and 4 =dentinal caries in the inner half of the dentine

ELIGIBILITY:
Inclusion Criteria:

* Extracted posterior teeth Visually intact occlusal surfaces or a variety of occlusal carious lesions, but no obvious cavities
* Removal of organic material and stains from the surfaces, the teeth will be immersed in 10% sodium hypochlorite solution for 20 min, followed by rinsing in distilled water for 20 min. The teeth will then stored in saturated thymol solution or formalin.
* The teeth will be arranged in pairs and mounted in plaster blocks.

Exclusion Criteria:

Teeth with deep cavity

-

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
To detect of occlusal caries | 4 months
  Primary Outcome Measure:
  1.To detect of occlusal caries To detect occlusal caries.42 teeth with initial non cavitated caries will be examined by kavodiagondent and then radiographed. The occlusal surfaces will be carefully scanned and measured 3 times when wet, and 3 times after they had been wiped with paper tissues and exposed to air for about 2 min in room temperature.the teeth will be radiographed.The radiographs will be examined by 4 radiologists. The observers will be instructed to select one of five ratings to represent his or her level of confidence that a carious lesion was present or not in the occlusal surfaces of the teeth. The following scale was used: 1 = definitely not caries, 2 = probably not Caries, 3 = questionable, 4 = probably caries, and 5 = definitely caries.
  the light microscope will be used as gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa Mahmoud elsayed, Cairo, Egypt